CLINICAL TRIAL: NCT01970176
Title: Define in Preclinical Systolic Dysfunction (PSD) With Renal Dysfunction, the Cardiorenal and Humoral Actions of Chronic Type V Phosphodiesterase (PDEV) Inhibition
Brief Title: Study to Determine How Cialis Effects the Renal Function in Response to Volume Expansion in Preclinical Systolic Cardiomyopathy (Aim2)
Acronym: Aim2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Horng Chen, MD, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 11-004644; HL76611-07P3 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cardiomyopathy; Renal Impairment
MeSH Terms: conditions — Cardiomyopathies; Renal Insufficiency | interventions — Tadalafil; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tadalafil (Active Comparator): Subject will receive Tadalafil daily for a total of 12 weeks
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Subject will receive Placebo daily for a total of 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil 5 mg tablet. Daily. Tadalafil dose varies from 5 mg to 20 mg for 12 weeks. If blood pressure is >95 then subject dismissed from the Clinical Research Unit (CRU) on 2 (5 mg) tabs of tadalafil or placebo. If blood pressure is between 90 - 95 mmHg systolic, then dismiss on 1 (5 mg) tab of Tadalafil. At 2 weeks (± 5 days) if blood pressure is> 100 than add 1 (5 mg) tab of Tadalafil to make a total of 3 (5mg) tabs of Tadalafil. At 4 weeks(± 5 days) if blood pressure is > 100 add 1 (5 mg) tab to make a total of 4 (5 mg) tablets of Tadalafil.
  Other Names: Tadalafil 5mg tablet
  Arms: Tadalafil
Drug: Placebo — Placebo tablet. Daily. Placebo tablets made to match appearance of 5mg Tadalafil tablets. Placebo dose varies from 5 mg to 20 mg (1 to 4 tablets) for 12 weeks. If blood pressure is >95 then subject dismissed from CRU on 2 tabs of placebo. If blood pressure is between 90 - 95 mmHg systolic, then dismiss on 1 (5 mg) tablet of placebo. At 2 weeks (± 5 days) if blood pressure is> 100 than add 1 tab of placebo to make a total of 3 tablets of placebo. At 4 weeks(± 5 days) if blood pressure is > 100 add 1 (5 mg) tab to make a total of 4 tablets of placebo.
  Other Names: Placebo tablet
  Arms: Placebo

SUMMARY:
To determine the effect of 12 weeks of chronic PDEV inhibition with Tadalafil versus placebo on basal cardiorenal and humoral function and on the integrated cardiorenal and humoral response to acute sodium loading in subjects with preclinical systolic dysfunction (PSD) and renal (kidney) dysfunction.

DETAILED DESCRIPTION:
At the consent visit a blood draw will be done also a the 6 minute walk will be done to determine eligibility and a physical exam along with vital signs, height and weight will be done. Twenty-four hour urine collection will be obtained one day prior to the active study day.

Prior to initiation of the study, subjects will be stabilized for at least one week on a no added salt diet (120 milliequivalents of sodium/salt per day (mEq Na/day) which will be maintained throughout the study period.

Subjects will be admitted to the Clinical Research Unit (CRU)on the evening before the active study day. They will be able to order a no-added salt meal and will not have anything to eat after midnight until the last renal clearance blood draw the next day. Bladder scan will be carried out to assess for urine retention. On the active study day, subjects take their medications upon awakening, however, diabetics will hold their diabetic medications until after the last renal clearance test then they will be able to order a regular diet meal and take their diabetic medications. Subjects will be asked to drink 5ml/Kg (milliliters per kilogram of body weight) of water to insure sufficient urinary flow. A priming dose (calculated according to body size) of Iothalamate, to measure glomerular filtration rate (GFR) and para-amino-hippurate (PAH) to measure effective renal plasma flow (ERPF) is infused, followed by a constant rate IV sustaining dose (calculated according to estimated kidney function) of Iothalamate or PAH. The subjects will be asked to empty their bladder spontaneously every thirty minutes. Throughout the study, at the end of each 30-minute clearance period, subjects will be asked to drink an amount of water equivalent to the sum of the blood losses and the urinary flow. After an equilibration period of 45 minutes, a 30-minute baseline renal clearance will be carried out.

Blood pressure will be measured at 20-minute intervals by using automatic blood pressure cuff, and heart rate will be continuously monitored by electrocardiography. Echocardiography will be performed during these baseline clearances to determine left atrial (LA) and Left Ventricular (LV)volumes and systolic and diastolic function.

After the baseline clearance the acute saline load will be administered (normal saline 0.9% 0.25 ml/kg/min for 1 hour). During the 1 hour saline load, one 30-minute clearance (as outlined above) will be repeated with the subjects in supine position after which a second 30-minute clearance will be repeated with the subject sitting or the head of the bed up. As above, blood samples are collected midway during each clearance and urine samples are obtained every 30 minutes. Echocardiography will be repeated immediately after the end of the saline infusion.

At the completion of the baseline renal clearance periods and response to acute sodium load, subjects will be randomized to Tadalafil or placebo. Subjects will be randomized in a 2:1 fashion.

All subjects will take oral Tadalafil (5 mg) or placebo once a day. The blood pressure will be checked prior to administering the drug.Thereafter, both blood pressure and heart rate will continue to be monitored for the next 4 hours. If after the first dose of study drug if patient's systolic blood pressure is < 85 mmHg systolic and has symptoms of hypotension e.g. lightheadedness, dizziness, feeling faint, blurred vision, the study drug will be stopped however the subject will continue in the study. After 2 hours if blood pressure is >95 systolic then give 1 more (5 mg) of Tadalafil or placebo and monitor blood pressure for 2 hours. If blood pressure is >95 then dismiss subject on 2 (5 mg) tabs of tadalafil or placebo. If blood pressure is between 90 - 95 mmHg systolic, then dismiss on 1 (5 mg) tab of Tadalafil or placebo.

Patients will then be dismissed. Subjects will also have access to a 24-hour phone number should they have any questions or develop any side effects. Subjects will return after one week (+ or - 4 days) for electrolyte check. They will also receive a weekly phone call to review status.

At 2 weeks (± 5 days) from dismissal if blood pressure is> 100 than add 1 (5 mg) tab of Tadalafil or placebo to make a total of 3 (5mg) tabs of Tadalafil or placebo.

At 4 weeks(± 5 days) if blood pressure is > 100 add 1 (5 mg) tab to make a total of 4 (5 mg) Tadalafil or placebo.

After six weeks( + or - 5 days) , subjects will repeat blood draw for safety labs (total blood count and electrolytes). For patients who do not live more than 25 miles away we will try to arrange this visit with the patient's local physician.

At the end of the twelve-week study period (+ or - 8 days), subjects will be admitted to the Clinical Research Unit the afternoon prior to the renal clearance study. Echocardiography, renal clearance, humoral determination and acute saline load will be performed in the same manner as the baseline study. Subjects will also perform a 24-hour urine collection the day prior to their return visit for determination of sodium excretion and creatinine clearance. Subjects will be dismissed after the renal clearance study.

ELIGIBILITY:
Inclusion Criteria:

* A total of 39 patients with PSD as defined by an ejection fraction of less than 40%, no clinical signs or symptoms of congestive heart failure, a minimal distance on 6-minute walk of equal or >450 meters will be recruited and calculated creatinine clearance of equal or less than 90 ml/min and greater than 30 ml/min, using the (MDRD-measurement of renal dysfunction, formula) assessed within the past 24 months. If the subject is not able to walk 450 meters due to pain in hips and knees and not fatigue or shortness of breath than they will still qualify for the protocol.

Exclusion Criteria:

* Current or anticipated future need for nitrate therapy

  * Systolic blood pressure < 90 mmHg or > 180 mm Hg
  * Diastolic blood pressure < 40 mmHg or > 100 mmHg
  * Patients taking alpha antagonists or cytochrome P450 3A4 inhibitors (ketoconazole, itraconazole, erythromycin, saquinavir, cimetidine or serum proteases inhibitors for HIV) who cannot be taken off these medications for the duration of the study.
  * Patients taking the following selective alpha blockers and who are unable to stop for the duration of the study;
  * Alfuzosin
  * Prazosin
  * Doxazosin
  * Tamsulosin
  * Terazosin
  * Silodosin
  * Patients with retinitis pigmentosa, previous diagnosis of nonischemic optic neuropathy, untreated proliferative retinopathy or unexplained visual disturbance
  * Patients with sickle cell anemia, multiple myeloma, leukemia or penile deformities placing them at risk for priapism (angulation, cavernosal fibrosis or Peyronie's disease)
  * Patients with an allergy to iodine.
  * Patients on PDEV inhibition for pulmonary hypertension
  * Patients on PDEV inhibition for erectile dysfunction who are not willing to stop the medication for the duration of the study
  * Valve disease (> moderate aortic or mitral stenosis; > moderate aortic or mitral regurgitation)
  * Obstructive Hypertrophic cardiomyopathy
  * Infiltrative or inflammatory myocardial disease (amyloid, sarcoid)
  * Pericardial disease
  * Have experienced a myocardial infarction or unstable angina, or have undergone percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) within 60 days prior to consent, or requires either PTCA or CABG at the time of consent
  * Severe congenital heart diseases
  * Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
  * Second or third degree heart block without a permanent cardiac pacemaker
  * Stroke within 3 months of screening or other evidence of significantly compromised Central Nervous System (CNS) perfusion
  * Hemoglobin <9 g/dL
  * Patients with severe liver disease (AST > 3x normal, alkaline phosphatase or bilirubin > 2x normal)
  * Serum sodium of < 125 mEq/dL or > 150 mEq/dL
  * Serum potassium of < 3.2 mEq/dL or > 5.9 mEq/dL
  * Prior diagnosis of intrinsic renal diseases including renal artery stenosis of > 50%
  * Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
  * Less than 21 years of age
  * Pregnant or nursing women.
  * Women of child bearing potential who do not have a negative pregnancy test at study entry and who are not using effective contraception
  * Non-cardiac condition limiting life expectancy to less than one year, per physician judgment
  * Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
  * Received an investigational drug within 1 month prior to dosing
  * In the opinion of the investigator is unlikely to comply with the study protocol or is unsuitable for any reasons

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H Chen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hubers SA, Wan SH, Adel FW, Benike SL, Burnett JC Jr, Scott C, Chen HH. Cardiorenal Effects of Long-Term Phosphodiesterase V Inhibition in Pre-Heart Failure. J Am Heart Assoc. 2022 Jan 18;11(2):e022126. doi: 10.1161/JAHA.121.022126. Epub 2022 Jan 8. PMID 35001638
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil: Subject received Tadalafil daily for a total of 12 weeks
  Tadalafil: Tadalafil 5 mg tablet. Daily. Tadalafil dose varies from 5 mg to 20 mg for 12 weeks. If blood pressure is >95 then subject dismissed from the Clinical Research Unit (CRU) on 2 (5 mg) tabs of tadalafil or placebo. If blood pressure is between 90 - 95 mmHg systolic, then dismiss on 1 (5 mg) tab of Tadalafil. At 2 weeks (± 5 days) if blood pressure is> 100 than add 1 (5 mg) tab of Tadalafil to make a total of 3 (5mg) tabs of Tadalafil. At 4 weeks(± 5 days) if blood pressure is > 100 add 1 (5 mg) tab to make a total of 4 (5 mg) tablets of Tadalafil.
- Placebo: Subject received Placebo daily for a total of 12 weeks
  Placebo: Placebo tablet. Daily. Placebo tablets made to match appearance of 5mg Tadalafil tablets. Placebo dose varies from 5 mg to 20 mg (1 to 4 tablets) for 12 weeks. If blood pressure is >95 then subject dismissed from CRU on 2 tabs of placebo. If blood pressure is between 90 - 95 mmHg systolic, then dismiss on 1 (5 mg) tablet of placebo. At 2 weeks (± 5 days) if blood pressure is> 100 than add 1 tab of placebo to make a total of 3 tablets of placebo. At 4 weeks(± 5 days) if blood pressure is > 100 add 1 (5 mg) tab to make a total of 4 tablets of placebo.
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 14 | 6
Completed | 14 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [58 to 73] | 64 [54 to 73] | 67 [56 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 6 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Sodium Excretion
Description: Change in total urinary sodium excretion as measured by MEq/min
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: MEq/min
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 14 | 6
MEq/min | 29.5 [-4.2 to 77.2] | 25.1 [2.9 to 61.3]
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Glomerular Filtration Rate (GFR)
Description: Change in total GFR as measured by ml/1.72m2
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: ml/1.72m2
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 14 | 6
ml/1.72m2 | -6.2 [-30.0 to -1.5] | 4.5 [-18.5 to 11]
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Urinary Cyclic Guanosine 3',5'-Monophosphate (cGMP) Hormone Excretion
Description: Change in total urinary cGMP hormone excretion as measured by pmol/min
Time Frame: Baseline, 12 weeks
Measure: Median (Inter-Quartile Range); unit: pmol/min
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 14 | 6
pmol/min | -71.1 [-266.0 to -41.0] | 51.6 [-198.0 to 237.0]
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 13 weeks.
Arm/Group | Tadalafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 8/14 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=14) | Placebo (N=6)
Indigestion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT01970176/Prot_SAP_000.pdf